CLINICAL TRIAL: NCT02528955
Title: De-intensification of Postoperative Radiotherapy in Selected Patients With Head and Neck Cancer
Brief Title: De-Intensification Radiotherapy Postoperative Head Neck
Acronym: DIREKHT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIREKHT
Record Dates: First submitted 2015-08-10; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Cancer of Head and Neck
Keywords: Head and neck cancer; postoperative; radiotherapy; de-intensification
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A:De-Intensification Radiotherapy (RT) primary tumor region (Active Comparator): A:De-Intensification Radiotherapy (RT) primary tumor region
  * ≤ pT2, R ≥ 5 mm, L0, Pn0
  * > 3 lymph node metastasis or patients with < 3 ipsilateral lymph node metastasis and a bilateral primary tumor without adequate contralateral neck dissection
  Interventions: Radiation: A: De-Intensification RT primary tumor region
- B:De-Intensification Radiotherapy contralateral lymph nodes (Active Comparator): * > pT2 and/or R < 5mm and/or L1 and/or Pn1
  * ≤ 3 ipsilateral lymph node metastasis (and contralateral pN0 (>= 6 resected lymph nodes) or contralateral cN0 in patients wih strictly ipsilateral localised ( >= 5 mm distance from midline) cancer of the oral cavity or oropharynx
  Interventions: Radiation: B: De-Intensification RT contralateral lymph nodes
- C:De-Intensification RT primary tumor region /contralateral LN (Active Comparator): * ≤ pT2, R ≥ 5 mm, L0, Pn0
  * ≤ 3 ipsilateral lymph node metastasis (and contralateral pN0 (>= 6 resected lymph nodes) or contralateral cN0 in patients wih strictly ipsilateral localised ( >= 5 mm distance from midline) cancer of the oral cavity or oropharynx
  Interventions: Radiation: C. De-Intensification RT primary tumor region AND contralateral lymph nodes

INTERVENTIONS:
Radiation: A: De-Intensification RT primary tumor region — A:
  * Reduction of radiation dose in the primary tumor region to 56 Gy,
  * Elective Radiotherapy of both neck sides
  Arms: A:De-Intensification Radiotherapy (RT) primary tumor region
Radiation: B: De-Intensification RT contralateral lymph nodes — B:
  * No dose reduction in primary tumor region (prescribed dose in primary tumor region: 64 Gy)
  * Reduction of target volume: only elective radiotherapy of the ipsilateral neck, no contralateral neck irradiation
  Arms: B:De-Intensification Radiotherapy contralateral lymph nodes
Radiation: C. De-Intensification RT primary tumor region AND contralateral lymph nodes — C:
  * Reduction of radiation dose in the primary tumor region to 56 Gy, AND
  * Reduction of target volume: only elective radiotherapy of the ipsilateral neck, no contralateral neck irradiation
  Arms: C:De-Intensification RT primary tumor region /contralateral LN

SUMMARY:
In patients with squamous cell carcinoma of the oral cavity, the oropharynx and larynx with >= pT3 and or pN+ postoperative radio - or radiochemotherapy is the standard of care. Postoperative radiochemotherapy is indicated in patients with multiple lymph node metastasis, lymph node metastasis with extracapsular spread and or R1/2 resection.

Locoregional control rates are over 80% after surgery and radio(chemo)therapy. But many patients suffer from therapy-related long-term side-effects, like xerostomia, dysphagia, fibrosis, trismus etc.

The aim of this study is to investigate if depending on primary tumor stage, quality of resection ( resection margin) and number of lymph node metastasis and performed neck dissection an adapted de-intensified dose- and target volume concept may be performed without reducing locoregional-control but with reducing radiotherapy-related side-effects.

DETAILED DESCRIPTION:
The study is a non-randomized phase-II trial. In total there are 3 therapy arms.

Patients are assigned to one of these therapy arms according to the tumor status and the quality and kind of surgery. The aim of this study is to investigate if a risk-adapted dose- and target-volume concept in clearly defined patient groups is possible to individualize postoperative radiotherapy without reducing locoregional-control but with reducing radiotherapy-related side-effects.

There are two main issues to investigate:

1. Dose prescription in primary tumor region:

   In this study it should be investigated if a dose reduction to 56 Gy in the primary tumor region is possible, if the resection margin is >= 5mm, tumor stage is <=pT2 and if there are no other risk factors like perineural spread or peritumoral lymphangiosis.
2. Target volume definition in elective lymph node levels

   It should be investigated if ipsilateral cervical lymph irradiation alone allows adequate locoregional control in selected patients:

   ipsilateral lymph node metastasis <=3 and contralateral pN0 (adequate contralateral selective neck dissection performed) or contralateral cN0 (in patients with strictly ipsilateral localized tumors of the oral cavity or oropharynx)

   Considering these facts 3 therapy groups are possible:

   A:

   Criteria:
   * pT2, R ≥ 5 mm, L0, Pn0

     * 3 lymph node metastasis or patients with < 3 ipsilateral lymph node metastasis and a bilateral primary tumor without adequate contralateral neck dissection

   Intervention:
   * Reduction of radiation dose in the primary tumor region to 56 Gy,
   * Elective Radiotherapy of both neck sides

   B:

   Criteria:

   •> pT2 and/or R < 5mm and/or L1 and/or Pn1

   •≤ 3 ipsilateral lymph node metastasis (and contralateral pN0 (>= 6 resected lymph nodes) or contralateral cN0 in patients wih strictly ipsilateral localised ( >= 5 mm distance from midline) cancer of the oral cavity or oropharynx

   Intervention

   •No dose reduction in primary tumor region (prescribed dose in primary tumor region: 64 Gy)

   •Reduction of target volume: only elective radiotherapy of the ipsilateral neck, no contralateral neck irradiation

   C:

   Criteria
   * pT2, R ≥ 5 mm, L0, Pn0
   * 3 ipsilateral lymph node metastasis (and contralateral pN0 (>= 6 resected lymph nodes) or contralateral cN0 in patients wih strictly ipsilateral localised ( >= 5 mm distance from midline) cancer of the oral cavity or oropharynx

   Intervention

   •Reduction of radiation dose in the primary tumor region to 56 Gy, AND

   •Reduction of target volume: only elective radiotherapy of the ipsilateral neck, no contralateral neck irradiation

   In all arms the dose prescription for the lymph node regions is as follows:

   •elective lymph node level (either ipsi- or bilateral): 50 Gy

   •lymph node level with lymph node metastasis without extracapsular extension: 56Gy
   * lymph node level with lymph node metastasis with extracapsular extension: 64 Gy

   In all arms simultaneously chemotherapy is recommended in the following cases:
   * lymph node metastasis with extracapsular extension •>= 3 lymph node metastasis

   All patients are stratified according to HPV status.

   Additional investigations:
   * swallowing endoscopy (before, 6 and 24 months after radiotherapy)
   * translational research (especially individual radiosensitivity, immunologic parameters in peripheral blood during treatment)
   * QoL

ELIGIBILITY:
Inclusion Criteria:

1. Histologic proven squamous cell carcinoma of the oral cavity/larynx/oro- or hypopharynx
2. Postoperative tumor status:

   * Oral cavity, oropharynx or larynx: pT1-3, pN0-pN2b
   * Hypopharynx: pT1-2; pN1
3. Patients that fulfill one or both of the following criteria:

   * ≤ pT2, R ≥ 5 mm, L0, Pn0
   * ≤ 3 ipsilateral lymph node metastases (if a contralateral adequate neck dissection is performed, no contralateral neck dissection is recommended in patients with strictly ipsilateral localised tumors of the oropharynx or oral cavity)
4. R0-Resection (resection margin ≥ 1mm)
5. No distant metastasis cM0
6. age ≥ 18 years, no upper age limit
7. ECOG ≤ 2
8. Patients that understood protocol contents and are able to behave according to protocol
9. Signed study-specific consent form prior to therapy
10. In case of indicated simultaneous chemotherapy:

    * adequate bone marrow function (leucocytes > 3,5x10^3, platelets > 100x 10^3, hemoglobin > 10g/dl
    * sufficient liver function: bilirubin < 2,0mg/dl, ALT, AST < less than 3 times upper limit of normal
    * sufficient renal function: normal serum creatinine, glomerular filtration rate > 60ml/min

Exclusion Criteria:

1. pregnant or lactating/nursing women
2. fertile patients that are not willing to use highly effective methods of contraception (per institutional standards) during treatment
3. Any condition potentially hampering compliance with the study protocol and follow-up schedule
4. On-treatment participation on other trials
5. R1 or R2 resection status
6. pN2c and pN3
7. cM1
8. prior radiotherapy in the head and neck region , prior chemo- or immunotherapy (neoadjuvant/induction)
9. time between surgery and beginning of radio(chemo)therapy > 6 weeks
10. Prior (> 4 months before beginning of radio(chemo)therapy) neck dissection
11. In case of indicated simultaneous chemotherapy:

    * reduced hearing ability (especially upper frequency range)
    * known dihydropyrimidindehydrogenase (DPD) deficiency
    * simultaneous therapy with brivudin or other DPD-inhibitors
    * uncontrolled serious disease, including physical and mental diseases, for example within last 6 months:instable angina pectoris, heart attack, serious cardiac dysrhythmias, stroke, serious carotid stenosis, neurologic or psychiatric disorders including epilepsy, dementia, psychosis; uncontrolled infection; liver cirrhosis Child B or C, severe hepatic impairment; severe blood count changes; severe renal impairment, HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-10; Primary Completion 2019-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
locoregional recurrence rate after 2 years | after 2 years
  (recurrence in-radiation field, radiation field margin, outside radiation field for example contralateral)

SECONDARY OUTCOMES:
Overall Survival | after 2 and 5 years
disease-free survival | after 2 and 5 years
distant-metastasis-free survival | after 2 and 5 years
acute toxicity according to ctc-ae v.4.0 | during therapy and up to 8 weeks after therapy
late toxicity according to ctc-ae v.4.0 | follow-up period (5years)
Quality of Life as measured by questionaires | before and during treatment and in the follow-up for 5 years
  questionaires: EORTC QLQ-C30 and QLQ-H&N35 and EAT-10

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Fietkau, Principal Investigator — Dept. of Radiooncology, University Hospital Erlangen
Locations (1):
- Dept. of Radiooncology, University Hospital, Erlangen, Germany

REFERENCES:
- [Derived] Haderlein M, Speer S, Ott O, Lettmaier S, Hecht M, Semrau S, Frey B, Scherl C, Iro H, Kesting M, Fietkau R. Dose Reduction to the Swallowing Apparatus and the Salivary Glands by De-Intensification of Postoperative Radiotherapy in Patients with Head and Neck Cancer: First (Treatment Planning) Results of the Prospective Multicenter DIREKHT Trial. Cancers (Basel). 2020 Feb 26;12(3):538. doi: 10.3390/cancers12030538. PMID 32110958
- [Derived] Onbasi Y, Lettmaier S, Hecht M, Semrau S, Iro H, Kesting M, Fietkau R, Haderlein M. Is there a patient population with squamous cell carcinoma of the head and neck region who might benefit from de-intensification of postoperative radiotherapy? : A monocentric retrospective analysis of a previously defined low-risk patient population treated with standard-of-care radiotherapy. Strahlenther Onkol. 2019 Jun;195(6):482-495. doi: 10.1007/s00066-018-1415-y. Epub 2019 Jan 4. PMID 30610355